CLINICAL TRIAL: NCT02627001
Title: Comparison of Air Leak During Ventilation With Nu-Mask Intraoral Airway Device Versus Conventional Bag Valve Mask in a Cadaver Model: A Randomized Crossover Trial
Brief Title: Nu-Mask Intraoral Airway Device Versus Conventional Bag Valve Mask Ventilation Crossover Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Program Director for Research, DEM, Brooke Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C.2014.134e
Record Dates: First submitted 2015-11-28; First posted 2015-12-10 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NuMask Intraoral Airway Device (Experimental): A United States Army Combat Medic uses a single hand technique to hold a Nu-Mask Intraoral Airway Device on a cadaver while an Impact 731 ventilator delivers 10 standardized breaths with tidal volumes of 750 ml each.
  Interventions: Device: NuMask Intraoral Airway Device
- Bag Valve Mask (Active Comparator): A United States Army Combat Medic uses a single hand technique to hold a conventional bag valve mask on a cadaver while an Impact 731 ventilator delivers 10 standardized breaths with tidal volumes of 750 ml each.
  Interventions: Device: Bag Valve Mask

INTERVENTIONS:
Device: NuMask Intraoral Airway Device — NuMask Intraoral Airway Device
  Arms: NuMask Intraoral Airway Device
Device: Bag Valve Mask — Conventional bag valve mask
  Arms: Bag Valve Mask

SUMMARY:
This study comprised a randomized cross-over trial of ventilation using the NuMask Intraoral Mask versus conventional Bag Valve Mask in a cadaver model among United States Army combat medics.

DETAILED DESCRIPTION:
This study comprised a randomized crossover trial of adult United States Army combat medic volunteers participating in a cadaver laboratory as part of their training. The study took place in Bulverde, TX. Participants were randomized to perform cadaver ventilation first using either the novel Nu-MaskR intraoral device or conventional bag valve mask. A one handed seal technique was used to simulate single operator ventilation. Participants were responsible for mask placement while a ventilator delivered 10 breaths each with a standardized tidal volume of 750 ml. After a 5-minute washout period, they performed ventilation using the alternative device. The primary outcome measure was air leak as calculated by subtracting tidal volume received from tidal volume delivered as measured by the ventilator.

ELIGIBILITY:
Inclusion Criteria:

* United States Army Combat Medics

Exclusion Criteria:

* Injuries precluding performance of bag valve mask ventilation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NuMask Intraoral Mask First, Then Standard Bag Valve Mask: A United States Army Combat Medic uses a single hand technique to hold a Nu-Mask Intraoral Airway Device on a cadaver while an Impact 731 ventilator delivers 10 standardized breaths with tidal volumes of 750 ml each. After a 5 minute rest period, the subject performs the same procedures using a conventional cuffed face mask.
  NuMask Intraoral Airway Device: NuMask Intraoral Airway Device
- Standard Bag Valve Mask First, Then Numask Intraoral Mask: A United States Army Combat Medic uses a single hand technique to hold a conventional bag valve mask on a cadaver while an Impact 731 ventilator delivers 10 standardized breaths with tidal volumes of 750 ml each. After a 5 minute rest period, the subject performs the same procedures using an intraoral mask.
  Bag Valve Mask: Conventional bag valve mask
Period: Overall Study
Arm/Group | NuMask Intraoral Mask First, Then Standard Bag Valve Mask | Standard Bag Valve Mask First, Then Numask Intraoral Mask
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NuMask Intraoral Mask First, Then Standard Bag Valve Mask: A United States Army Combat Medic uses a single hand technique to hold a Nu-Mask Intraoral Airway Device on a cadaver while an Impact 731 ventilator delivers 10 standardized breaths with tidal volumes of 750 ml each. The Medic then performs the same procedures using a standard bag valve mask.
  NuMask Intraoral Airway Device: NuMask Intraoral Airway Device
- Standard Bag Valve Mask First, Then Numask Intraoral Mask: A United States Army Combat Medic uses a single hand technique to hold a conventional bag valve mask on a cadaver while an Impact 731 ventilator delivers 10 standardized breaths with tidal volumes of 750 ml each. The Medic then performs the same procedures using a Nu-Mask Intraoral Airway Device.
  Bag Valve Mask: Conventional bag valve mask
- Total: Total of all reporting groups
Arm/Group | NuMask Intraoral Mask First, Then Standard Bag Valve Mask | Standard Bag Valve Mask First, Then Numask Intraoral Mask | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 013 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Received Minute Volume (Liters) as Measured by Wright Respirometer
Description: An Impact 731 Ventilator will be attached to a mask. Subjects will hold a mask seal on a cadaver for 100 seconds. The Impact 731 Ventilator will then deliver standardized tidal volumes of 750 cc (delivered tidal volume) 10 times at six second intervals. A Wright respirometer will then measure received tidal volume for each of these 10 breaths.
Time Frame: 1 Minute
Measure: Median (Inter-Quartile Range); unit: Liters
Arm/Group | NuMask Intraoral Airway Device | Bag Valve Mask
Number analyzed (Participants) | 27 | 27
Liters | 6.8 [5.7 to 7.2] | 5.2 [4.4 to 6.3]
Statistical Analysis 1: Comparison: NuMask Intraoral Airway Device vs Bag Valve Mask; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Ranks

ADVERSE EVENTS:
Arm/Group | NuMask Intraoral Airway Device | Bag Valve Mask
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No